CLINICAL TRIAL: NCT06278818
Title: Neural and Clinical Correlates of Rehabilitation in Neurodegenerative Conditions
Brief Title: Effects of Telerehabilitation on Brain Network Connectivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: University of Parma (Other); University of Bologna (Other); University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MNESYS-PE0000006
Record Dates: First submitted 2024-02-06; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Non-pharmacological treatments; Cognitive training; Rehabilitation; Dementia; Connectivity; Neuroimaging
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The neurophysiologist and neuroradiologist will be blinded to the type of rehabilitation treatment (experimental group vs. control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Network-based Cognitive Training (NBCT) (Experimental): The training will be delivered through a virtual platform for TR.
  Interventions: Behavioral: Cognitive Telerehabilitation
- Home-based Cognitive Rehabilitation (HomeCoRe) (Experimental): The training will be delivered through a touch-screen laptop in a home-based setting.
  Interventions: Behavioral: Cognitive Telerehabilitation
- Semantic Memory Rehabilitation Training (SMRT) (Experimental): The training will be delivered through TR with the assistance of an online therapist.
  Interventions: Behavioral: Cognitive Telerehabilitation
- Unstructured Home-based Cognitive Stimulation (Control) (Sham Comparator): The Control stimulation will be delivered through TR with therapist assistance.
  Interventions: Other: Control Condition

INTERVENTIONS:
Behavioral: Cognitive Telerehabilitation — Cognitive training specifically designed to promote cognitive functions in early stages of neurodegenerative conditions.
  Arms: Home-based Cognitive Rehabilitation (HomeCoRe); Network-based Cognitive Training (NBCT); Semantic Memory Rehabilitation Training (SMRT)
Other: Control Condition — This activity is commonly used as a control condition to test the effectiveness of innovative rehabilitative treatments.
  Arms: Unstructured Home-based Cognitive Stimulation (Control)

SUMMARY:
The current project aims at assessing the impact of various cognitive telerehabilitation approaches on patients with Mild Cognitive Impairment (MCI) associated with neurodegenerative diseases, namely Alzheimer's disease (AD) and Parkinson's disease (PD). The study focuses on non-pharmacological interventions to maintain patients' residual functionality, limit disease progression, and improve quality of life for both patients and their caregivers.

This longitudinal and multicenter study applies innovative cognitive telerehabilitation (TR) methods and evaluates their impact on functional parameters obtained with high-density electroencephalogram (HD-EEG) and resting-state functional magnetic resonance imaging (rsFMRI). The goal is to identify neurophysiological correlates of the effects of three different cognitive TR in individuals with MCI due to neurodegenerative conditions.

The study aims to:

* Identify correlations between improvement in cognitive performance and functional brain data.
* Use acquired knowledge to develop neurologically guided TR approaches for broader use.

The research will include patients diagnosed with MCI associated with neurodegenerative diseases. Primary outcome measures include changes in resting-state brain connectivity assessed through HD-EEG and rsFMRI. Secondary outcomes involve the assessment of changes in neuropsychological measures, caregiver burden, immediately after rehabilitation and after longitudinal follow-up.

The study is designed to last 30 months, with follow-up assessments at three time points. The primary outcomes will be evaluated using rsFMRI and HD-EEG instrumental acquisitions, the secondary outcomes will be evaluated using clinical assessments and neuropsychological tests.

DETAILED DESCRIPTION:
Currently, the impact of drug therapies on neurodegenerative conditions is very limited; The drugs available are mostly symptomatic and recent drug trials with new molecules have given contrasting results about the possibility of slowing down progression of disease. Therefore, clinically there is a strong interest in possible non-pharmacological intervention strategies for preserving functionality and limiting progression of disease as far as possible, reducing disability, and improving quality of life for both patients and their caregivers. Neurodegenerative diseases, such as Alzheimer's disease (AD) and, in some cases Parkinson's disease (PD), are characterized by a progressive cognitive decline. During the initial and mild cognitive impairment (MCI) phase, subjects report subjective disorders and show an objective and measurable cognitive impairment, although they maintain independence in day-to-day life activities. No consensus has been reached on the effect of non-pharmacological approaches to contrast cognitive decline, but there is a general agreement that these approaches are more likely to succeed the sooner they are implemented and the more accurately they act on the domains involved in the cognitive decline process.

The current longitudinal and multicenter study aims to apply innovative cognitive telerehabilitation (TR) approaches to the MCI population, to assess the impact of the different cognitive telerehabilitation approaches on brain network connectivity, acquired by means of high-density electroencephalogram (HD-EEG) and functional magnetic resonance imaging at rest (rs-fMRI). Moreover, the protocol will evaluate the effects of cognitive TR on neuropsychological measures. The primary outcome will be evaluated by means of a direct comparison between brain network connectivity measures before and after the intervention and by means of a comparison with a control group of MCI subjects, who will be involved in unstructured cognitive activities.

Condition Condition: Early stages of cognitive impairment due to neurodegenerative diseases, i.e. AD and PD.

Telerehabilitation Approaches Network-based Cognitive Training (NBCT) - A cognitive training specifically designed to promote the co-activation of multiple brain areas (i.e., central nodes), modulating the functional connectivity of specific resting state networks (RSNs) (i.e., Default Mode Network, DMN, e Salience Network, SN). This rehabilitation package has been used in face-to-face mode on a sample of healthy subjects (average age: 66 years), in whom a rehabilitation-induced "up-regulation" effect of the functional connectivity of the rear central nodes of the DMN was observed. Subsequently, this training approach has been tested in MCI-AD, MCI-PD and in patients with relapsing-remitting multiple sclerosis who complained of mild cognitive deficits. Within the framework of this study, the rehabilitation program will be implemented on a telerehabilitation platform (i.e. Khymeia) and will be administered through a virtual connection. A link will be provided for each rehabilitation session, which will allow participants to access and use the rehabilitation protocol through a web browser on their personal computer, tablet or mobile. This approach offers many advantages in terms of practicality, ease of use and accessibility for study participants.

Home-based Cognitive Rehabilitation (HomeCoRe) system - software for cognitive rehabilitation specially developed for the initial stages of deterioration (amnestic MCI, MCI-PD, mild AD), the usability and effectiveness of both in the person version (CoRe), as well as in remote rehabilitation (HomeCore) in the short and long term has been verified in the hospital field also in combination with neurostimulation techniques. HomeCoRe is an adaptive patient-tailored treatment that returns a Weighted score of performance for each exercise and each session to monitor patient's progress even remotely and adjust the level of difficulty of the proposed exercises accordingly. The mentioned strategy is applied to avoid over or under stimulation of the patient. The software provides an easy to access platform through which the patient interacts via a touch screen. The usability and acceptance of the home version of HomeCoRe has already been tested in a small group of patients in the early stages of cognitive impairment.

Semantic Memory Rehabilitation Training (SMRT) - Building upon the crucial role that the processing of semantic aspects of episodic information plays in long-term episodic memory processes, and recent evidence indicating early involvement of semantic memory in preclinical forms of Alzheimer's disease, the current cognitive training aims to enhance semantic processing in patients with MCI. The dual objective is to improve both episodic and semantic memory processes. A pilot study has yielded encouraging results in a small group of patients. The protocol is administered through telerehabilitation using a specific device with constant assistance from an online therapist.

Unstructured Home-based Cognitive Stimulation (Control) - This activity is commonly used as a control condition to test the effectiveness of innovative rehabilitative treatments, such as NBTC, HomeCoRe, and SMRT in this case. The treatment involves 60 minutes of daily activities (frequency and overall treatment duration will be adapted to the experimental treatment for comparison). Patients will receive instructions from the therapist along with a participant diary. For each session, few newspaper articles will be provided for the patient to read and summarize in the diary by answering specific questions. The protocol is administered through tele-rehabilitation using a specific device with constant assistance from an online therapist.

ELIGIBILITY:
Inclusion criteria for MCI-AD subjects:

* Confirmed clinical diagnosis of MCI due to possible Alzheimer's disease with evidence of AD pathophysiological processes, according to National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association criteria (Albert et al., 2011);
* Ability to understand and consciously sign informed consent and adhere to study procedures.
* Educational level ≥ 5 years.

Inclusion criteria for MCI-PD subjects:

* Clinical diagnosis of MCI-PD according to Level II criteria (Litvan et al., 2012). Ability to understand and consciously sign informed consent and adhere to study procedures.
* Educational level ≥ 5 years.

Exclusion criteria:

* Aphasia, visuospatial neglect;
* Atypical and/or secondary parkinsonisms;
* Dementia according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria;
* Alterations of consciousness;
* Sensory disorders that could interfere with the execution of tests and rehabilitative treatment;
* Concurrent psychiatric and/or neurological and/or essential tremor disorders;
* Presence of systemic inflammatory and infectious diseases, autoimmune diseases, malignant tumors at the time of recruitment, deemed clinically significant by the investigator and therefore capable of interfering with the study results;
* Inability or unwillingness to undergo MRI and/or EEG;
* Presence of prostheses or metallic implants incompatible with MRI;
* Deep brain stimulation (DBS) implant.
* Any dropouts will be managed by enrolling new patients.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in resting-state brain networks functional connectivity after NBTC treatment | Between-session before (Week 0) - after (Week 4 +/-2) NBCT TR
  Change in the resting-state functional connectivity from Baseline (T0) to the end of NBCT TR (T1 after 4 weeks) as measured by rs-fMRI. Connectivity measures will be extracted by means of Independent Component Analysis (ICA) and seed-based connectivity analysis approaches. This approach allowed for a detailed exploration of the functional connectivity networks associated with potential effects of NBTC treatment.
Changes in resting-state EEG coherence after NBTC treatment | Between-session before (Week 0) - after (Week 4 +/-2) NBCT TR
  Change in the resting-state coherence from Baseline (T0) to the end of NBCT TR (T1 after 4 weeks) as measured by HD-EEG. Connectivity measures will be extracted by means of seed-based connectivity analysis. This approach allowed for a detailed exploration of the HD-EEG connectivity networks associated with potential effects of NBTC treatment.
Changes in resting-state EEG coherence after HomeCore treatment | Between-session before (Week 0) - after (Week 6 +/-2) HomeCore TR
  Change in the resting-state coherence from Baseline (T0) to the end of HomeCore TR (T1 after 6 weeks) as measured by HD-EEG. Connectivity measures will be extracted by means of seed-based connectivity analysis. This approach allowed for a detailed exploration of the HD-EEG connectivity networks associated with potential effects of HomeCore treatment.
Changes in resting-state brain networks functional connectivity after SMRT treatment | Between-session before (Week 0) - after (Week 6 +/-2) SMRT TR
  Change in the resting-state functional connectivity from Baseline (T0) to the end of SMRT TR (T1 after 6 weeks) as measured by rs-fMRI. Connectivity measures will be extracted by means of Independent Component Analysis (ICA) and seed-based connectivity analysis approaches. This approach allowed for a detailed exploration of the functional connectivity networks associated with potential effects of SMRT treatment.

SECONDARY OUTCOMES:
Changes in neuropsychological and caregiver burden measures after TR | Between-session TO (Week 0) - T1 (Week 4 +/-2 or 6 +/-2) - T2 (Week 30+/-2 or 32+/-2) - T3 (Week 56+/-2 or 58+/-2)
  The efficacy of TR will be assessed by comparing neuropsychological tests and caregiver burden measures obtained across evaluation sessions (T0-T3). Changes in neuropsychological and caregiver burden measures will be correlated with the strength of changes in rs-fMRI or HD-EEG brain connectivity obtained comparing T0 to T1.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, Principal Investigator — University of Pavia
Locations (1):
- IRCCS Mondino Foundation, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publication of the study protocol.
Supporting Information: Study Protocol
Time Frame: The data will be available after acceptance of the study protocol by the Open Access Journal.
Access Criteria: Paper download.

REFERENCES:
- [Background] Wright LM, De Marco M, Venneri A. Verbal fluency discrepancies as a marker of the prehippocampal stages of Alzheimer's disease. Neuropsychology. 2023 Oct;37(7):790-800. doi: 10.1037/neu0000836. Epub 2022 Jun 23. PMID 35737533
- [Background] Rodella C, Bernini S, Panzarasa S, Sinforiani E, Picascia M, Quaglini S, Cavallini E, Vecchi T, Tassorelli C, Bottiroli S. A double-blind randomized controlled trial combining cognitive training (CoRe) and neurostimulation (tDCS) in the early stages of cognitive impairment. Aging Clin Exp Res. 2022 Jan;34(1):73-83. doi: 10.1007/s40520-021-01912-0. Epub 2021 Jun 22. PMID 34156651
- [Background] Quaglini S, Panzarasa S, Alloni A, Sacchi M, Sinforiani E, Bottiroli S, Bernini S. HomeCoRe: Bringing Cognitive Rehabilitation at Home. Stud Health Technol Inform. 2019 Aug 21;264:1755-1756. doi: 10.3233/SHTI190632. PMID 31438328
- [Background] Manca R, Mitolo M, Wilkinson ID, Paling D, Sharrack B, Venneri A. A network-based cognitive training induces cognitive improvements and neuroplastic changes in patients with relapsing-remitting multiple sclerosis: an exploratory case-control study. Neural Regen Res. 2021 Jun;16(6):1111-1120. doi: 10.4103/1673-5374.300450. PMID 33269758
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] De Marco M, Venneri A. Volume and Connectivity of the Ventral Tegmental Area are Linked to Neurocognitive Signatures of Alzheimer's Disease in Humans. J Alzheimers Dis. 2018;63(1):167-180. doi: 10.3233/JAD-171018. PMID 29578486
- [Background] De Marco M, Meneghello F, Duzzi D, Rigon J, Pilosio C, Venneri A. Cognitive stimulation of the default-mode network modulates functional connectivity in healthy aging. Brain Res Bull. 2016 Mar;121:26-41. doi: 10.1016/j.brainresbull.2015.12.001. Epub 2015 Dec 11. PMID 26688237
- [Background] Bernini S, Stasolla F, Panzarasa S, Quaglini S, Sinforiani E, Sandrini G, Vecchi T, Tassorelli C, Bottiroli S. Cognitive Telerehabilitation for Older Adults With Neurodegenerative Diseases in the COVID-19 Era: A Perspective Study. Front Neurol. 2021 Jan 14;11:623933. doi: 10.3389/fneur.2020.623933. eCollection 2020. PMID 33519704
- [Background] Bernini S, Panzarasa S, Sinforiani E, Quaglini S, Cappa SF, Cerami C, Tassorelli C, Vecchi T, Bottiroli S. HomeCoRe for Telerehabilitation in Mild or Major Neurocognitive Disorders: A Study Protocol for a Randomized Controlled Trial. Front Neurol. 2021 Dec 23;12:752830. doi: 10.3389/fneur.2021.752830. eCollection 2021. PMID 35002919
- [Background] Bernini S, Ballante E, Fassio F, Panzarasa S, Quaglini S, Riccietti C, Costa A, Cappa SF, Tassorelli C, Vecchi T, Bottiroli S. In person versus remote cognitive rehabilitation in patients with subjective cognitive decline or neurocognitive disorders: what factors drive patient's preference? Front Psychol. 2023 Oct 4;14:1266314. doi: 10.3389/fpsyg.2023.1266314. eCollection 2023. PMID 37868592
- [Background] Bernini S, Panzarasa S, Barbieri M, Sinforiani E, Quaglini S, Tassorelli C, Bottiroli S. A double-blind randomized controlled trial of the efficacy of cognitive training delivered using two different methods in mild cognitive impairment in Parkinson's disease: preliminary report of benefits associated with the use of a computerized tool. Aging Clin Exp Res. 2021 Jun;33(6):1567-1575. doi: 10.1007/s40520-020-01665-2. Epub 2020 Sep 8. PMID 32895890
- [Background] Bernini S, Gerbasi A, Panzarasa S, Quaglini S, Ramusino MC, Costa A, Avenali M, Tassorelli C, Vecchi T, Bottiroli S. Outcomes of a computer-based cognitive training (CoRe) in early phases of cognitive decline: a data-driven cluster analysis. Sci Rep. 2023 Feb 7;13(1):2175. doi: 10.1038/s41598-022-26924-2. PMID 36750612
- [Background] Bernini S, Alloni A, Panzarasa S, Picascia M, Quaglini S, Tassorelli C, Sinforiani E. A computer-based cognitive training in Mild Cognitive Impairment in Parkinson's Disease. NeuroRehabilitation. 2019;44(4):555-567. doi: 10.3233/NRE-192714. PMID 31256092
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Derived] Caminiti SP, Bernini S, Bottiroli S, Mitolo M, Manca R, Grillo V, Avenali M, De Icco R, Capellari S, Carlesimo GA, Venneri A, Tassorelli C. Exploring the neural and behavioral correlates of cognitive telerehabilitation in mild cognitive impairment with three distinct approaches. Front Aging Neurosci. 2024 Jun 27;16:1425784. doi: 10.3389/fnagi.2024.1425784. eCollection 2024. PMID 38993694